CLINICAL TRIAL: NCT01040078
Title: Novel Influenza A/H1N1 Split- Virion Vaccine in Healthy Children Aged 6 to 35 Month
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Xiaofeng Liang
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 20090601
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 7.5ug H1N1 vaccine (Experimental): 360 subjects to receive two doses 7.5ug H1N1 influenza vaccine on Day 0 and Day 21.
  Interventions: Biological: 7.5ug H1N1 Influenza vaccine
- 15ug H1N1 vaccine (Experimental): 360 subjects to receive two doses 15ug H1N1 influenza vaccine on Day 0 and Day 21.
  Interventions: Biological: 15ug H1N1 vaccine
- seasonal influenza vaccine (Placebo Comparator): 180 subjects to receive two doses seasonal influenza vaccine on Day 0 and Day 21.
  Interventions: Biological: seasonal influenza vaccine

INTERVENTIONS:
Biological: 7.5ug H1N1 Influenza vaccine — 0.25 mL intramuscular injection into the deltoid region of the arm on Day 0 and day 21
  Arms: 7.5ug H1N1 vaccine
Biological: 15ug H1N1 vaccine — 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and day 21
  Arms: 15ug H1N1 vaccine
Biological: seasonal influenza vaccine — 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and day 21
  Arms: seasonal influenza vaccine

SUMMARY:
The purpose of this study is to generate data on immunogenicity and safety of the monovalent H1N1 vaccine in support of the development and registration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >= 6 months to =<35 months at the time of the first study vaccination. Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative Subject and parent/legal representative are able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months which might interfere with the assessment of immune response
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia contraindicating intramuscular (IM) vaccination as reported by parents/legal representative
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Chronic illness that in the opinion of the Investigator is at a stage where it might interfere with trial conduct or completion
* Family members of the employees or the Investigator
* Previous participation in a trial investigating a vaccine with the swine-origin A/H1N1 influenza strain
* Confirmed infection with the novel influenza A/H1N1 strain
* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-02 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Lingchuan County CDC, Guilin, Guangxi
  - Luxi County CDC, Xiangxi Prefecture, Hunan
  - Yandu District CDC, Yancheng, Jiangsu